CLINICAL TRIAL: NCT00274950
Title: Protocol for the Treatment of Extracranial Germ Cell Tumours in Children and Adolescents (GC III)
Brief Title: Observation and/or Combination Chemotherapy After Surgery or Biopsy in Treating Young Patients With Extracranial Germ Cell Tumors
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Children's Cancer and Leukaemia Group (Other)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000454553; CCLG-GC-2005-04; EUDRACT-2004-002503-33; EU-20584
Record Dates: First submitted 2006-01-10; First posted 2006-01-11 (Estimated); Last update posted 2013-09-17 (Estimated); Status verified 2009-06

CONDITIONS: Childhood Germ Cell Tumor; Extragonadal Germ Cell Tumor; Ovarian Cancer
Keywords: childhood extragonadal germ cell tumor; childhood malignant ovarian germ cell tumor; childhood malignant testicular germ cell tumor; recurrent childhood malignant germ cell tumor; childhood teratoma; childhood extracranial germ cell tumor
MeSH Terms: conditions — Ovarian Neoplasms; Ovarian Germ Cell Cancer; Testicular Neoplasms; Teratoma | interventions — Bleomycin; Carboplatin; Cisplatin; Etoposide; Ifosfamide; Vinblastine; Chemotherapy, Adjuvant

INTERVENTIONS:
Biological: bleomycin sulfate
Drug: carboplatin
Drug: cisplatin
Drug: etoposide
Drug: ifosfamide
Drug: vinblastine sulfate
Procedure: adjuvant therapy
Procedure: conventional surgery

SUMMARY:
RATIONALE: Sometimes, after surgery, the tumor may not need additional treatment until it progresses. In this case, observation may be sufficient. Drugs used in chemotherapy work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more tumor cells. Giving combination chemotherapy after surgery may kill any remaining tumor cells.

PURPOSE: This phase III trial is studying how well observation and/or combination chemotherapy works after surgery or biopsy in treating young patients with extracranial germ cell tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

* Stratify and reduce treatment for pediatric patients with extracranial germ cell tumors while maintaining event-free survival.
* Treat newly diagnosed patients with extracranial germ cell tumors requiring chemotherapy with a carboplatin-based strategy.
* Develop a common strategy for the treatment of patients with recurrent or progressive extracranial germ cell tumors.
* Register all cases of mature and immature teratoma.
* Develop a common strategy for the management of immature and mature teratoma, including follow-up strategies to permit early detection of yolk sac recurrence.

OUTLINE: This is a multicenter study.

Patients who have not had prior biopsy or surgical resection undergo biopsy (if feasible) or surgical resection. Patients with mature or immature teratoma undergo observation. These patients who relapse (i.e., tumor regrowth) may undergo further surgical resection unless tumor markers are significantly elevated. If the tumor markers are significantly elevated, these patients proceed to JEB chemotherapy according to risk group. Patients with all other malignant germ cell tumors are assigned to 1 of 3 treatment groups according to risk.

* Low-risk group: Patients with normal tumor markers undergo observation. Patients with rising tumor markers only AND no imageable tumor proceed to treatment as in the intermediate-risk group. Patients with rising tumor markers AND/OR imageable tumor are considered to have relapsed and proceed to treatment as in the intermediate- or high-risk group.
* Intermediate-risk group: Patients receive JEB chemotherapy comprising etoposide IV over 4 hours on days 1-3, carboplatin IV over 1 hour on day 2, and bleomycin IV over 30 minutes on day 3. Treatment repeats every 21 days for 4 courses. Patients with residual tumors after completion of chemotherapy may undergo second-look surgery.
* High-risk group: Patients receive JEB chemotherapy as in the intermediate-risk group for 6 courses. Patients with residual tumors after completion of chemotherapy may undergo second-look surgery.
* Relapse therapy: Patients in the intermediate- or high-risk group who relapse after completion of JEB chemotherapy receive vinblastine IV on days 1 and 2, ifosfamide IV over 1 hour on days 1-5, and cisplatin IV on days 1-5. Treatment repeats every 21 days for 6 courses.

PROJECTED ACCRUAL: A total of 105 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically* proven extracranial malignant germ cell tumor (GCT), including mature/immature teratoma, with or without elevated alpha-fetoprotein (AFP) or human chorionic gonadotropin (HCG) levels

  * Newly diagnosed disease
  * Patients with relapsed or progressive extracranial malignant GCT allowed if previously treated with carboplatin, etoposide, and bleomycin (JEB) chemotherapy

    * Patients relapsing following JEB are eligible for the study relapse strategy NOTE: *Patients with unequivocally raised AFP/HCG whose risk of biopsy is felt to be high can be diagnosed by clinical grounds, imaging, and markers
* No intracranial GCTs

PATIENT CHARACTERISTICS:

* Neutrophil count ≥ 1,000/mm^3
* Platelet count ≥ 100,000/mm^3
* Bilirubin ≤ 2 times upper limit of normal (ULN)
* ALT ≤ 3 times ULN
* Not pregnant or nursing

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior chemotherapy other than JEB

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 105 (Estimated)
Dates: Start 2005-05; Primary Completion 2010-05 (Estimated)

PRIMARY OUTCOMES:
Event-free survival
Continuation of treatment
Development of common and follow-up strategies
Registration of all cases of mature and immature teratoma

CONTACTS AND LOCATIONS:
Overall Officials: Juliet Hale, MD, Principal Investigator — Sir James Spence Institute of Child Health at Royal Victoria Infirmary
Locations (20):
- Our Lady's Hospital for Sick Children Crumlin, Dublin, Ireland
- United Kingdom (19):
  - Birmingham Children's Hospital, Birmingham, England
  - Institute of Child Health at University of Bristol, Bristol, England
  - Addenbrooke's Hospital, Cambridge, England
  - Leeds Cancer Centre at St. James's University Hospital, Leeds, England
  - Leicester Royal Infirmary, Leicester, England
  - Royal Liverpool Children's Hospital, Alder Hey, Liverpool, England
  - Royal London Hospital, London, England
  - Great Ormond Street Hospital for Children, London, England
  - Royal Manchester Children's Hospital, Manchester, England
  - Sir James Spence Institute of Child Health at Royal Victoria Infirmary, Newcastle upon Tyne, England
  - Queen's Medical Centre, Nottingham, England
  - Children's Hospital - Sheffield, Sheffield, England
  - Southampton General Hospital, Southampton, England
  - Royal Marsden - Surrey, Sutton, England
  - Royal Belfast Hospital for Sick Children, Belfast, Northern Ireland
  - Royal Aberdeen Children's Hospital, Aberdeen, Scotland
  - Royal Hospital for Sick Children, Edinburgh, Scotland
  - Royal Hospital for Sick Children, Glasgow, Scotland
  - Childrens Hospital for Wales, Cardiff, Wales